CLINICAL TRIAL: NCT02191735
Title: Performance Evaluation of the RAMP® Cardiac Tests / RAMP® 200 in a Point-Of-Care Setting (C-POC)
Brief Title: RAMP 200 / RAMP Cardiovascular Tests at the Point-of-Care
Acronym: C-POC
Status: Completed | Type: Observational
Sponsor: Response Biomedical Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP024
Record Dates: First submitted 2014-07-10; First posted 2014-07-16 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Heart Failure; Congestive Heart Failure
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — EDTA plamsa specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Troponin I: Subjects who have undergone a routine test order of Troponin for suspected Acute Coronary Syndrome / Myocardial Infarction (ACS/MI). Waste sample blood will then be tested on the RAMP 200 and the RAMP Reader for comparison.
  Interventions: Device: RAMP 200; Device: RAMP Reader
- Myoglobin: Subjects who have undergone a routine test order of Troponin for suspected Acute Coronary Syndrome / Myocardial Infarction (ACS/MI) and who have a RAMP Myoglobin test result that is within the test reportable range. Waste sample blood will then be tested on the RAMP 200 and the RAMP Reader for comparison.
  Interventions: Device: RAMP 200; Device: RAMP Reader
- CK-MB: Subjects who have undergone a routine test order of Troponin for suspected Acute Coronary Syndrome / Myocardial Infarction (ACS/MI) and who have a RAMP CK-MB test result that is within the test reportable range. Waste sample blood will then be tested on the RAMP 200 and the RAMP Reader for comparison.
  Interventions: Device: RAMP 200; Device: RAMP Reader
- NT-proBNP: Subjects who have undergone a routine test order of NT-proBNP or BNP for suspected Heart Failure (HF). Waste sample blood will then be tested on the RAMP 200 and the RAMP Reader for comparison.
  Interventions: Device: RAMP 200; Device: RAMP Reader

INTERVENTIONS:
Device: RAMP 200 — The RAMP® Reader is a general use fluorometer that analyzes results produced by immunoassays that use a fluorophore having an excitation wavelength at 560 nm and an emission wavelength of 610 nm. The RAMP® 200 is Response Biomedical's second generation reader. The RAMP® 200 is designed to process more tests with a smaller footprint.
Device: RAMP Reader — The RAMP® Reader is a general use fluorometer that analyzes results produced by immunoassays that use a fluorophore having an excitation wavelength at 560 nm and an emission wavelength of 610 nm. The RAMP® Reader is Response Biomedical's first generation reader instrument. Designed for use at near-patient/bedside or locations such as: laboratories, hospitals, on-site Emergency Response and Emergency Rooms.

SUMMARY:
This clinical investigation is designed to demonstrate the performance characteristics of the RAMP® cardiac tests analyzed on the RAMP® 200 by non-laboratorial Operators at the point-of-care when compared to the results for the same samples analyzed on the RAMP® Reader.

ELIGIBILITY:
Inclusion Criteria:

Study Arms A - Troponin I (ACS/MI)

1. Males or Females, 18 years of age or older, of any race
2. Has had a routine test order of Troponin for suspected Acute Coronary Syndrome / Myocardial Infarction (ACS/MI) - as per institutional guidelines
3. Willing to voluntarily agree to sign a consent form (if applicable)

Study Arms B - Myoglobin (ACS/MI)

1. Males or Females, 18 years of age or older, of any race
2. Has had a routine test order of Troponin for suspected Acute Coronary Syndrome / Myocardial Infarction (ACS/MI) - as per institutional guidelines
3. Myoglobin test result falls within the reportable range of the test as reported in the RAMP® Myoglobin IFU.
4. Willing to voluntarily agree to sign a consent form (if applicable)

Study Arms C - CK-MB (ACS/MI)

1. Males or Females, 18 years of age or older, of any race
2. Has had a routine test order of Troponin for suspected Acute Coronary Syndrome / Myocardial Infarction (ACS/MI) - as per institutional guidelines
3. CK-MB test result falls within the reportable range of the test as reported in the RAMP® CK-MB IFU.
4. Willing to voluntarily agree to sign a consent form (if applicable)

Study Arm D - NT-proBNP (HF)

1. Males or Females, 18 years of age or older, of any race
2. Has had a routine test order of NT-proBNP or BNP for suspected Heart Failure (HF) - as per institutional guidelines
3. Willing to voluntarily agree to sign a consent form (if applicable)

Exclusion Criteria:

Study Arms A, B, C - Troponin I, Myoglobin, CK-MB (ACS/MI)

1. Healthy Subjects
2. Pregnant or lactating
3. Subjects not having a cardiac marker test ordered
4. Blood sample collected >24 hours prior to screening
5. Subjects without adequate volumes of surplus EDTA whole blood available for all required trial testing
6. Non-compliance to the protocol or the inclusion criteria

Study Arm D - NT-proBNP (HF)

1. Healthy Subjects
2. Pregnant or lactating
3. Subjects not having a cardiac marker test ordered
4. Blood sample collected >24 hours prior to screening
5. Subjects without adequate volumes of surplus EDTA whole blood available for all required trial testing
6. Non-compliance to the protocol or the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 600 total subjects, 18 years of age and older will be enrolled into this study at a minimum of 3 sites in the United States of America (USA).
  Each site will screen for a minimum of approximately 200 clinical surplus whole blood samples derived from subjects presenting with symptoms and signs indicative of cardiovascular heart disease (i.e. acute myocardial infarction and/or heart failure). It is expected that the population will be divided approximately equally between males and females. Clinical site enrollment will be monitored throughout the trial to verify population distribution.
Sampling Method: Non-Probability Sample
Enrollment: 719 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Substantial Equivalence of the RAMP® Reader and the RAMP® 200 when running the RAMP® Cardiac tests. | method comparison - subjects will be followed for the duration of 1 blood draw, with a total study enrollment over 3 months.
  The primary objective is to achieve substantial equivalence of the RAMP® cardiac tests on the RAMP® Reader and the RAMP® 200 in a point-of-care (POC) setting by evaluating the following analytical performance specifications:
  * precision on the RAMP® 200, when used at maximum complexity, utilizing frozen control materials;
  * precision on the RAMP® 200, when used at maximum complexity, utilizing whole blood specimens; and,
  * performance via method comparison across the reportable ranges of the RAMP® cardiac tests.

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Christenson, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (3):
- United States (3):
  - San Francisco General Hospital, San Francisco, California
  - University of Maryland Medical Center, Baltimore, Maryland
  - Minneapolis Medical Research Foundation, Minneapolis, Minnesota